CLINICAL TRIAL: NCT04819646
Title: An Open-label, Single-arm Study to Evaluate the Effects of a Marine Lipid Oil Concentrate Formulation on Inflammation/Discomfort in Individuals Who Are Generally Healthy
Brief Title: Evaluate the Effects of a Marine Lipid Oil Concentrate Formulation on Inflammation/Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Supplement Formulators, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CL108
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Inflammation
Keywords: inflammation; Pain; Discomfort; Soreness
MeSH Terms: conditions — Inflammation; Pain | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inflammation (Experimental): Marine Lipid Oil concentrate softgel and dietary supplement capsule
  Interventions: Dietary Supplement: Marine Lipid Oil Concentrate Formulation; Dietary Supplement: Dietary Supplement

INTERVENTIONS:
Dietary Supplement: Marine Lipid Oil Concentrate Formulation — Marine Lipid Oil Concentrate softgels
Dietary Supplement: Dietary Supplement — Dietary Supplement capsules

SUMMARY:
The purpose of the study is to assess the efficacy and safety of a Marine Lipid Oil Concentrate formulation on inflammation/discomfort and overall well-being in male and female subjects who are generally healthy

DETAILED DESCRIPTION:
This is an open-label, single-arm remote study to evaluate the effects of a Marine Lipid Oil Concentrate formulation on inflammation/discomfort and overall well-being in individuals who are generally healthy. Each subject will receive a specific dose of the study products to be taken once daily for a total of 60 days.

Participants complete assessments and questionnaires.

The primary objective is the evaluation of the change in the responses to the SF-36 (Short-Form-36) Health Survey, Medical Symptoms questionnaire, Pain questionnaire and responses on an assessment form relative to baseline.

Safety and tolerability will be evaluated through receipt of documentation and responses from the telephone contacts/emails as per protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory, male or female, 35-75 years of age
2. Indicating "very mild," "mild, "or "moderate" for question #7 on the SF-36 Health Survey (How much bodily pain have you had during the past 4 weeks?)
3. Have had minor body discomfort, pain, or soreness occurring at least four times per week during the past 4 weeks including symptoms felt when arising in the morning, at the end of a day, during or after physical activity
4. Have personal access and able to operate a smartphone, tablet, or computer with enough memory to accommodate additional application(s) and have a reliable internet service
5. Able to print out and return documents by scan, email or by mail
6. Generally healthy and having no significant difficulty with digestion or absorption of food
7. Able to complete an Activity Log and Study Product Log daily
8. Has been generally weight stable for the past six months (+/- 6 lbs.)
9. Willing and able to give written informed consent
10. Clearly understands the procedures and study requirements
11. Willing and able to comply with all study procedures, including following recommendations to maintain their usual diet and regular activity, as per protocol
12. Able to communicate, including reading, in English
13. Has not taken any nutritional supplements that may contain any of the components of the study products for a minimum of 14 days before Screening/baseline and for the duration of the study period -

Exclusion Criteria:

1. Not having basic skills needed to operate a smartphone, tablet, or computer
2. Having smoked any cigarette, electronic cigarette, cigar, pipe, or used a recreational drug as well as any product containing cannabidiol (CBD) and tetrahydrocannabinol (THC) in the past 30 days
3. Having donated blood within 30 days before Screening/baseline
4. Having been diagnosed with dysphagia or difficulty swallowing
5. Having participated in another study within 30 days prior to Screening/baseline
6. Being pregnant or planning on becoming pregnant during study participation; or breast feeding
7. History of allergy or sensitivity to any component of the study products
8. Having taken a lipid lowering medication (including statin medications) on a consistent basis for > 3 months and have muscle-related pain and/or anticipate a change in the medication during the study period
9. Currently taking a medication or dietary supplement specifically for pain or inflammation, including curcumin, and unwilling to washout (i.e., stop taking medication or supplement) for 14 days before Screening/baseline
10. Currently taking or having taken a fish oil, krill oil, omega-3 supplement and omega-3 prescription drugs within the past 3 months before Screening/baseline which, in the judgment of the Study Investigator/Sub-Investigator, would preclude participation in study
11. Currently taking or having taken pain medications or anti-inflammatory medication(s) (e.g., aspirin > 325 mg, non-steroidal anti-inflammatory drugs [NSAIDs], COX-2 (Cyclooxygenase-2) inhibitors, and corticosteroids) within 14 days before Screening/baseline which, in the judgment of the Study Investigator/Sub-Investigator would preclude participation in the study
12. Having been diagnosed, received medical treatment, or taking medication daily for the following medical condition(s):

    * Acute or chronic inflammatory or autoimmune disease (including rheumatoid arthritis, systemic lupus erythematosus, ankylosing spondylitis, Sjögren's syndrome, polymyalgia rheumatica, inflammatory bowel disease, and psoriatic arthritis)
    * Active infection
    * Active periodontal disease
13. Having been in an accident or had surgery with resulting body discomfort, pain, or soreness
14. Having been diagnosed with a pain-related disorder or under the care of a pain specialist
15. Presence of active or recurring clinically significant conditions as follows:

    * Diabetes mellitus or other endocrine disease
    * Eating disorder
    * Cardiovascular disease including heart and blood vessel disease, arrhythmia, heart attack, stroke, or heart valve problem
    * Gastrointestinal disease including gallbladder problems, gallstones, or biliary tract obstruction
    * Thyroid disease (unless on a stable dose of medication for ≥ 3 months before Screening/baseline and unlikely to change medication or dose during the study)
    * Hypertension (unless on a stable dose of medication for ≥ 3 months before Screening/baseline and unlikely to change medication or dose during the study)
    * Neurologic condition/disease
    * Cancer (unless skin cancer other than melanoma which has been treated ≥ 3 years before Screening/baseline)
    * Liver, pancreatic, and kidney disease
    * Pulmonary disease
    * Blood coagulation disorder or other hematologic disease
    * Other condition or medication use that would preclude participation in the study in the judgment of the Study Investigator/Sub-Investigator
16. Currently taking any medication or treatment for a psychiatric disorder (bipolar disorder, manic disorder, schizophrenia, apathetic [inherited] disorder), that include antidepressant drugs, including selective serotonin reuptake inhibitors (SSRIs), tricyclic and atypical antidepressants; benzodiazepines; phenothiazines, central nervous system (CNS) depressants as well as the following medications: dextromethorphan, meperidine, monoamine oxidase inhibitors (MAOIs), pentazocine and tramadol. These may preclude participation in the study dependent on the judgment of the Study Investigator/Sub-Investigator.
17. Currently taking or having taken within the 30 days before Screening/baseline any hormone replacement therapy (including DHEA (dehydroepiandrosterone), estrogen, progesterone, or testosterone), except those utilized as a method of birth control and which have been taken for > 3 months with no anticipated change for the duration of the study period
18. Having had a surgical procedure or having an internal medical device which, in the judgment of the Study Investigator/Sub-Investigator, would preclude participation in the study
19. Currently consumes more than 7 standard alcoholic drinks per week for women and 4 drinks per week for men (a standard alcoholic drink is defined as one bottle/can of beer, one glass of wine, or one ounce of hard liquor)
20. Unable or unwilling to avoid consuming grapefruit juice or fresh grapefruit, Seville oranges, and tangelos for the duration of the study period
21. History of known or suspected substance abuse (e.g., alcohol, opiates, benzodiazepines or amphetamines)
22. Having any other circumstance that precludes study participation in the judgment of the Study Investigator/Sub-Investigator, including use of other nutritional supplements, which will be evaluated on a case-by-case basis

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
SF-36 (Short Form-36) Health Survey | 60 days
  Assessment of the mean change in the results from the SF-36 Health Survey from baseline
Medical Symptoms Questionnaire | 60 days
  Assessment of the mean change in the results from the Medical Symptoms Questionnaire from baseline
Pain Questionnaire | 60 days
  Assessment of the mean change in the results from the Pain Questionnaire from baseline
Minor body discomfort, pain, or soreness | 60 days
  Assessment of the mean change in the frequency of minor body discomfort, pain, or soreness per week from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Swick, Ph.D, Principal Investigator — Life Extension
Locations (1):
- Lfie Extension Clinical Reseach, Inc., Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aggarwal BB, Gupta SC, Sung B. Curcumin: an orally bioavailable blocker of TNF and other pro-inflammatory biomarkers. Br J Pharmacol. 2013 Aug;169(8):1672-92. doi: 10.1111/bph.12131. PMID 23425071
- [Background] Bassiouny AR, Zaky A, Kandeel KM. Alteration of AP-endonuclease1 expression in curcumin-treated fibrotic rats. Ann Hepatol. 2011 Oct-Dec;10(4):516-30. PMID 21911894
- [Background] Buhrmann C, Mobasheri A, Busch F, Aldinger C, Stahlmann R, Montaseri A, Shakibaei M. Curcumin modulates nuclear factor kappaB (NF-kappaB)-mediated inflammation in human tenocytes in vitro: role of the phosphatidylinositol 3-kinase/Akt pathway. J Biol Chem. 2011 Aug 12;286(32):28556-66. doi: 10.1074/jbc.M111.256180. Epub 2011 Jun 13. PMID 21669872
- [Background] Campbell, M., Berrones, A., Krishnakumar, I. M., Charnigo, R. J., Westgate, P. M., & Fleenor, B. S. (2017). Responsiveness to curcumin intervention is associated with reduced aortic stiffness in young, obese men with higher initial stiffness. J Funct Foods, 29, 154-160.
- [Background] Campbell MS, Ouyang A, I M K, Charnigo RJ, Westgate PM, Fleenor BS. Influence of enhanced bioavailable curcumin on obesity-associated cardiovascular disease risk factors and arterial function: A double-blinded, randomized, controlled trial. Nutrition. 2019 Jun;62:135-139. doi: 10.1016/j.nut.2019.01.002. Epub 2019 Jan 11. PMID 30889454
- [Background] Chainani-Wu N, Madden E, Lozada-Nur F, Silverman S Jr. High-dose curcuminoids are efficacious in the reduction in symptoms and signs of oral lichen planus. J Am Acad Dermatol. 2012 May;66(5):752-60. doi: 10.1016/j.jaad.2011.04.022. Epub 2011 Sep 9. PMID 21907450
- [Background] Chen FY, Zhou J, Guo N, Ma WG, Huang X, Wang H, Yuan ZY. Curcumin retunes cholesterol transport homeostasis and inflammation response in M1 macrophage to prevent atherosclerosis. Biochem Biophys Res Commun. 2015 Nov 27;467(4):872-8. doi: 10.1016/j.bbrc.2015.10.051. Epub 2015 Oct 19. PMID 26471308
- [Background] Doyle R, Sadlier DM, Godson C. Pro-resolving lipid mediators: Agents of anti-ageing? Semin Immunol. 2018 Dec;40:36-48. doi: 10.1016/j.smim.2018.09.002. Epub 2018 Oct 4. PMID 30293857
- [Background] Fiala M, Terrando N, Dalli J. Specialized Pro-Resolving Mediators from Omega-3 Fatty Acids Improve Amyloid-beta Phagocytosis and Regulate Inflammation in Patients with Minor Cognitive Impairment. J Alzheimers Dis. 2015;48(2):293-301. doi: 10.3233/JAD-150367. PMID 26401996
- [Background] Hewlings SJ, Kalman DS. Curcumin: A Review of Its Effects on Human Health. Foods. 2017 Oct 22;6(10):92. doi: 10.3390/foods6100092. PMID 29065496
- [Background] Krishnakumar, I. M., Abhilash, M., Gopakumar, G., Dinesh, K., Balu, M., & Ramadasan, K. (2015). Improved blood-brain-barrier permeability and tissue distribution following the oral administration of a food-grade formulation of curcumin with fenugreek fibre. J Funct Foods, 14, 215-225.
- [Background] T Krishnareddy N, Thomas JV, Nair SS, N Mulakal J, Maliakel BP, Krishnakumar IM. A Novel Curcumin-Galactomannoside Complex Delivery System Improves Hepatic Function Markers in Chronic Alcoholics: A Double-Blinded, randomized, Placebo-Controlled Study. Biomed Res Int. 2018 Sep 23;2018:9159281. doi: 10.1155/2018/9159281. eCollection 2018. PMID 30345312
- [Background] Kumar, D., Jacob, D., Subash, P. S., Abhilash, M., Johannah, N. M., Ramadassan, K., . Krishnakumar, I. M. (2016). Enhanced bioavailability and relative distribution of free (unconjugated) curcuminoids following the oral administration of a food-grade formulation with fenugreek dietary fibre: A randomised double-blind crossover study. J Funct Foods, 22, 578 - 587.
- [Background] Lopez-Vicario C, Rius B, Alcaraz-Quiles J, Garcia-Alonso V, Lopategi A, Titos E, Claria J. Pro-resolving mediators produced from EPA and DHA: Overview of the pathways involved and their mechanisms in metabolic syndrome and related liver diseases. Eur J Pharmacol. 2016 Aug 15;785:133-143. doi: 10.1016/j.ejphar.2015.03.092. Epub 2015 May 15. PMID 25987424
- [Background] Madhu K, Chanda K, Saji MJ. Safety and efficacy of Curcuma longa extract in the treatment of painful knee osteoarthritis: a randomized placebo-controlled trial. Inflammopharmacology. 2013 Apr;21(2):129-36. doi: 10.1007/s10787-012-0163-3. Epub 2012 Dec 16. PMID 23242572
- [Background] Mehra MR, Lavie CJ, Ventura HO, Milani RV. Fish oils produce anti-inflammatory effects and improve body weight in severe heart failure. J Heart Lung Transplant. 2006 Jul;25(7):834-8. doi: 10.1016/j.healun.2006.03.005. Epub 2006 May 24. PMID 16818127
- [Background] Menon VP, Sudheer AR. Antioxidant and anti-inflammatory properties of curcumin. Adv Exp Med Biol. 2007;595:105-25. doi: 10.1007/978-0-387-46401-5_3. PMID 17569207
- [Background] Nathan C, Ding A. Nonresolving inflammation. Cell. 2010 Mar 19;140(6):871-82. doi: 10.1016/j.cell.2010.02.029. PMID 20303877
- [Background] Nordgren TM, Anderson Berry A, Van Ormer M, Zoucha S, Elliott E, Johnson R, McGinn E, Cave C, Rilett K, Weishaar K, Maddipati SS, Appeah H, Hanson C. Omega-3 Fatty Acid Supplementation, Pro-Resolving Mediators, and Clinical Outcomes in Maternal-Infant Pairs. Nutrients. 2019 Jan 5;11(1):98. doi: 10.3390/nu11010098. PMID 30621269
- [Background] Norling LV, Ly L, Dalli J. Resolving inflammation by using nutrition therapy: roles for specialized proresolving mediators. Curr Opin Clin Nutr Metab Care. 2017 Mar;20(2):145-152. doi: 10.1097/MCO.0000000000000353. PMID 28002074
- [Background] Norris PC, Skulas-Ray AC, Riley I, Richter CK, Kris-Etherton PM, Jensen GL, Serhan CN, Maddipati KR. Identification of specialized pro-resolving mediator clusters from healthy adults after intravenous low-dose endotoxin and omega-3 supplementation: a methodological validation. Sci Rep. 2018 Dec 21;8(1):18050. doi: 10.1038/s41598-018-36679-4. PMID 30575798
- [Background] Panahi Y, Hosseini MS, Khalili N, Naimi E, Simental-Mendia LE, Majeed M, Sahebkar A. Effects of curcumin on serum cytokine concentrations in subjects with metabolic syndrome: A post-hoc analysis of a randomized controlled trial. Biomed Pharmacother. 2016 Aug;82:578-82. doi: 10.1016/j.biopha.2016.05.037. Epub 2016 Jun 6. PMID 27470399
- [Background] Saji S, Asha S, Svenia PJ, Ratheesh M, Sheethal S, Sandya S, Krishnakumar IM. Curcumin-galactomannoside complex inhibits pathogenesis in Ox-LDL-challenged human peripheral blood mononuclear cells. Inflammopharmacology. 2018 Oct;26(5):1273-1282. doi: 10.1007/s10787-018-0474-0. Epub 2018 Apr 9. PMID 29633105
- [Background] Serhan CN. Discovery of specialized pro-resolving mediators marks the dawn of resolution physiology and pharmacology. Mol Aspects Med. 2017 Dec;58:1-11. doi: 10.1016/j.mam.2017.03.001. Epub 2017 Mar 3. PMID 28263773
- [Background] So J, Wu D, Lichtenstein AH, Tai AK, Matthan NR, Maddipati KR, Lamon-Fava S. EPA and DHA differentially modulate monocyte inflammatory response in subjects with chronic inflammation in part via plasma specialized pro-resolving lipid mediators: A randomized, double-blind, crossover study. Atherosclerosis. 2021 Jan;316:90-98. doi: 10.1016/j.atherosclerosis.2020.11.018. Epub 2020 Dec 7. PMID 33303222
- [Background] Spite M, Claria J, Serhan CN. Resolvins, specialized proresolving lipid mediators, and their potential roles in metabolic diseases. Cell Metab. 2014 Jan 7;19(1):21-36. doi: 10.1016/j.cmet.2013.10.006. Epub 2013 Nov 14. PMID 24239568
- [Background] Wongcharoen W, Jai-Aue S, Phrommintikul A, Nawarawong W, Woragidpoonpol S, Tepsuwan T, Sukonthasarn A, Apaijai N, Chattipakorn N. Effects of curcuminoids on frequency of acute myocardial infarction after coronary artery bypass grafting. Am J Cardiol. 2012 Jul 1;110(1):40-4. doi: 10.1016/j.amjcard.2012.02.043. Epub 2012 Apr 3. PMID 22481014
- [Background] Yu Y, Shen Q, Lai Y, Park SY, Ou X, Lin D, Jin M, Zhang W. Anti-inflammatory Effects of Curcumin in Microglial Cells. Front Pharmacol. 2018 Apr 20;9:386. doi: 10.3389/fphar.2018.00386. eCollection 2018. PMID 29731715